CLINICAL TRIAL: NCT07163390
Title: Iron Deficiency Anemia in the Second and Third Trimester of Pregnancy: Evaluation of the Contribution of Sucrosomial Iron Supplementation (Sideral® Folico)
Brief Title: Iron Deficiency Anemia in the Second and Third Trimester of Pregnancy
Acronym: PESO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 7816
Record Dates: First submitted 2025-08-25; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Anemia, Iron Deficiency; Pregnancy Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iron deficiency anemia in pregnancy (Experimental): Women with ongoing pregnancy attending at Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome will be prospectively enrolled from 24 to 32 weeks of pregnancy whether their hemoglobin levels are comprised between 8.5 and 10.5 g/dl. Patients will discontinue any other ongoing oral supplementation.
  Interventions: Combination Product: Sideral Folico

INTERVENTIONS:
Combination Product: Sideral Folico — Pregnant women will be enrolled from 24 to 32 weeks of gestation whether their hemoglobin levels are comprised between 8.5 and 10.5 g/dl. They start oral supplementation with Sucrosomial iron® 30 mg (Sideral® Folico), 2 sticks for twice a day for 15 days, followed by Sucrosomial iron ® 30 mg (Sideral® Folico), 1 stick for twice a day for the next 15 days

SUMMARY:
Iron deficiency is the most frequent cause of anemia during pregnancy and of maternal blood transfusion during the post-partum period. Intravenous administration is the fastest route to correct iron deficiency, bypassing the filter of iron intestinal absorption, the only true mechanism of iron balance regulation in the human body. Intravenous iron administration is suggested in patients who are refractory/intolerant to oral iron sulfate. This approach is expected to increase of at least 1 gr/dL the level of hemoglobin in 4 weeks. However, the intravenous route of iron administration has some drawbacks; first it is allowed only as in-hospital procedure and requires a resuscitation service, in accordance with the recommendations of the European Medicine Agency. Moreover, it is very expensive and negatively affects patient's perceived quality of life. A new oral iron formulation, Sucrosomial iron, bypassing the normal route of absorption, appears to be better tolerated and more cost-effective in correcting iron deficiency anemia at doses higher than those usually effective with other oral iron formulations. The hypothesis of the present study is that oral sucrosomial iron can correct iron deficiency anemia during pregnancy comparably to intravenous ferrous sulphate, with less side effects.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women from 24 to 32 weeks of pregnancy
* Age ≥18 ys old
* Hemoglobin between 8.5 and 10.5 g/dl
* Ability to sign an informed written consent

Exclusion Criteria:

* Patients with preclampsia
* twin pregnancy
* chronic diseases
* drug exposure
* BMI<18 or >30
* malabsorption
* fetal growth restriction
* age < 18 years
* haematologic diseases
* symptomatic anemia (dyspnea, tachycardia)
* inability to sign an informed written consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Anemia correction | one month
  to evaluate the contribution of the product Sucrosomial iron® 30 mg (Sideral® Folico) to determine a rise of 1g/dl of haemoglobin in 30 days of supplementation. To this end the patients will undergo to the following exams:
  - T0: evaluation of blood levels of Hb, Ferritin, sideremia, mean globular volume (MCV), transferrin saturation, Reactive C-Protein (PCR), according to routine clinical practice. Collection of medical and obstetric history and anthropometric parameters. Record of red meat consumption (more or less than twice a week).
  These evaluations will be made after after 15 days from the beginning of the supplementation, according to routine clinical practice (T1) and after 30 days from the beginning of the supplementation (T2)

SECONDARY OUTCOMES:
Compliance of treatment | 15 days
  to evaluate the tolerability of the product Sucrosomial iron® 30 mg (Sideral® Folico) the Visual Analogue Scale (VAS) or the 0-10 numeric scale for gastrointestinal pain will be used. Other assessments include measuring the rate of nausea, constipation or diarrhea, and dark or black stools. All evaluations will be made at T0, T1 and T2.

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Paradisi, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS